CLINICAL TRIAL: NCT06389903
Title: Study of Symptoms Related to the Lesion Effect Associated With the Implantation of Electrodes for Stimulation of the Subthalamic Nuclei in the Treatment of Parkinson's Disease.
Brief Title: Subthalamic Nucleus Stimulation Electrode and Psychiatric Lesion Effects in Parkinson's Disease
Acronym: PSYLES-STIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier du Rouvray (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-A00185-50
Record Dates: First submitted 2023-10-06; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease
Keywords: Brain stimulation
MeSH Terms: conditions — Parkinson Disease | interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavorial Assessment (Experimental): post-surgery behavioral assessment using scales
  Interventions: Behavioral: assessment

INTERVENTIONS:
Behavioral: assessment — post-surgery behavioral assessment using scales

SUMMARY:
This is a pilot, prospective, monocentric study concerning 15 Parkinson's disease patients requiring deep brain stimulation implantation.

The primary objective is to evaluate the psychiatric lesion effects of deep brain stimulation in patients with Parkinson's disease, using the Young Mania Rating Scale (YMRS), Big Five Inventory and the Hamilton Depression Rating Scale (HAMD 21).

DETAILED DESCRIPTION:
The patients included were adults suffering from Parkinson's disease (according to ICD-10). They had no severe psychiatric disorders, and no major neurocognitive disorders contraindicating surgery. An initial evaluation will be carried out 72 hours after surgery, then after one month, and finally 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Diagnosis of Parkinson's disease (ICD-10)
* L-dopa test must be positive
* Participants who gave their informed, written consent

Exclusion Criteria:

* Severe psychiatric disorder
* Major neurocognitive disorder contraindicating surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2020-07-03 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
Assessment of change of mania symptoms | Baseline, 72 hours, 1 month and 3 months after surgery
  The variation of Young Mania Rating Scale (YMRS). The YMRS total score ranges from 0 to 60 where higher scores indicate more severe mania.

SECONDARY OUTCOMES:
Assessment of change of depressive symptoms | Baseline, 72 hours, 1 month and 3 months after surgery
  The variation of Hamilton Rating Scale for Depression (HAMD-21). HAMD21 is a 21-item assessment used to measure depression severity. Items were rated on a scale from 0 (symptoms not present) to a maximum of 2 to 4 (symptom extremely severe) for a total score ranging from 0 (not at all depressed) to 64 (severely depressed).
Assessment of change of Behavior | Baseline, 72 hours, 1 month and 3 months after surgery
  The variation of the Ardouin Scale of Behavior in Parkinson's Disease. The total score ranges from 0 to 84. Higher score mean worse outcome.
Assessment of change of Impulsivity | Baseline, 72 hours, 1 month and 3 months after surgery
  The variation of the Dickman Impulsivity Inventory. It is a self report measure assessing dysfunctional impulsivity and functional impulsivity. Regarding dysfunctional impulsivity (12 items), higher score mean worse adaptation. Regarding functional impulsivity (11 items), higher score mean better adaptation.
Assessment of change of Apathy | Baseline, 72 hours, 1 month and 3 months after surgery
  The variation of the Apathy Evaluation Scale. This 18 item scale ranges from 0 to 12. Higher score means worse outcome.
Assessment of personality | Baseline
  Big Five inventory. The test identified five factors as follows :
  * openness to experience (inventive/curious vs. consistent/cautious)
  * conscientiousness (efficient/organized vs. extravagant/careless)
  * extraversion (outgoing/energetic vs. solitary/reserved)
  * agreeableness (friendly/compassionate vs. critical/judgmental)
  * neuroticism (sensitive/nervous vs. resilient/confident)
Assessment of executive functions | Baseline, 72 hours, 3 months after surgery
  Frontal Assessment Battery at Bedside. Thebattery consists of six subtests exploring the following: conceptualization, mental flexibility, motor programming, sensitivity to interference, inhibitory control, and environmental autonomy.
Assessment of confusion | 72 hours and 3 months after surgery
  Confusion Assessment method (CAM). The CAM instrument assesses the presence, severity, and fluctuation of 9 delirium features: acute onset, inattention, disorganized thinking, altered level of consciousness, disorientation, memory impairment, perceptual disturbances, psychomotor agitation or retardation, and altered sleep-wake cycle.

CONTACTS AND LOCATIONS:
Locations (1):
- Marie Desbordes, MD, Sotteville-lès-Rouen, France

IPD SHARING:
Plan to Share IPD: No